CLINICAL TRIAL: NCT03333239
Title: Short-term, Long-term and Cost-effectiveness of Treating Depression and Anxiety Disorders in Children and Adolescents - a Randomized Controlled Trial
Brief Title: Short-term, Long-term and Cost-effectiveness of Treating Depression and Anxiety Disorders in Children and Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University of Bremen (Other)
Responsible Party: Principal Investigator, Silke Wiegand-Grefe, Prof. Dr., Prof. Dr., Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: vakjp_2
Record Dates: First submitted 2017-09-04; First posted 2017-11-06 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Depression, Anxiety
Keywords: childhood and adolescence
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Psychotherapy, Psychodynamic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- psychodynamic psychotherapy (Experimental)
  Interventions: Behavioral: psychodynamic psychotherapy
- cognitive behavioral psychotherapy (Experimental)
  Interventions: Behavioral: cognitive behavioral psychotherapy
- psychodynamic family intervention (Active Comparator)
  Interventions: Behavioral: psychodynamic family intervention

INTERVENTIONS:
Behavioral: psychodynamic psychotherapy — the intervention follows the published in german manual: Psychoanalytische Behandlung von Kindern und Jugendlichen mit Angststörungen und Depressionen: Behandlungsmanual (Baumeister-Duru, Hofmann, Timmermann & Wulf, 2013)
  Arms: psychodynamic psychotherapy
Behavioral: cognitive behavioral psychotherapy — the interventions follow the published in german manuals: Depression (Ihle, Groen, Walter, Esser, & Petermann, 2012) and Soziale Ängste und Leistungsängste (Büch, Döpfner, & Petermann, 2015)
  Arms: cognitive behavioral psychotherapy
Behavioral: psychodynamic family intervention — the intervention follows an adapted version of the manual: Chimp´s - Children of mentally ill parents (Wiegand-Gefe, Halverscheid, & Plass, 2011)
  Arms: psychodynamic family intervention

SUMMARY:
The current study will evaluate and compare the effectiveness of cognitive-behavioral and psychodynamic therapy. Therefore 420 children and adolescents (ages 8-16 years) with depression and/or anxiety disorder will be randomly assigned to a treatment or a control condition. The intervention´s short-term effectiveness and sustainability as well as cost-effectiveness will be examined over a 5 year period for each participant.

DETAILED DESCRIPTION:
This study aims to optimize patient-centered care and to ensure scientific and legal approval of cognitive-behavioral and psychodynamic therapy for children and adolescents in the German health-care system. This prospective, randomized and controlled trial will therefore compare psychodynamic and cognitive behavioral therapy with a low-frequency family intervention (control intervention) for children and adolescents with depression and anxiety disorder. Number of diagnoses or fulfilled diagnostic criteria - diagnosed by a trained psychologist who is blind for treatment condition - will be the primary outcome. Secondary outcomes are patients´ and parents´ strain caused by symptoms, patients´ quality of life, global and family functioning and treatments´ cost effectiveness are secondary outcomes.

Patients will be recruited at the end of an inpatient hospital stay in northern Germany (Hamburg and Bremen) in two clinics for child and adolescent psychiatry and in surgery. After gathering informed consent from parents and patients, the latter will be randomly assigned to one type of outpatient treatment (psychodynamic, cognitive behavioral therapy or family intervention). Psychodynamic and cognitive-behavioral therapy as well as the control intervention will be provided manual-based. Treatment sessions will be audio recorded to control adherence.

Data will be collected annually over a period of five years starting at the beginning of treatment. This allows examination of varying treatment intervals as well as the sustainability and health economics of therapy effects.

To analyze data, comparisons of means will be performed. Groupwise analyses of interaction will be performed for inferential testing of differences in subgroups. Differences in therapy effects will be inferentially analyzed by multifactor analysis of covariance, analysis of variance or logistic regression. Interaction effects and predicting variables are of special interest.

In a Subsample of 32 depressive adolescents (ages 13-16) patients expectations before and experiences whilst therapy will be analyzed by a mixed-methods-approach.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of a depressive disorder (ICD-10; F30-F39) or an anxiety disorder (ICD-10; F40-F42)
* informed consent
* ages 8 to 16 years

Exclusion Criteria:

* psychotic disorders, eating disorders, substance use related disorders (except caffeine and nicotine), autism spectrum disorders, mutism, personality disorders
* neurologic disorders
* severe mental retardation (filling out questionnaires and interview are not feasible)
* low command of the german language

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Estimated)
Dates: Start 2017-12-22 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline children´s psychiatric symptomatology at 12 months | baseline and 12 months
  Children´s psychiatric symptomatology will be assessed in all groups (intervention groups and control group) by an external independent interview (Kiddie-SADS; Kaufman et al., 1996). The Kiddie-SADS interview will be conducted by a trained rater external to the project.
Change from baseline children´s psychiatric symptomatology at 24 months | baseline and 24 months
  Children´s psychiatric symptomatology will be assessed in all groups (intervention groups and control group) by an external independent interview (Kiddie-SADS; Kaufman et al., 1996). The Kiddie-SADS interview will be conducted by a trained rater external to the project.
Change from baseline children´s psychiatric symptomatology at 36 months | baseline and 36 months
  Children´s psychiatric symptomatology will be assessed in all groups (intervention groups and control group) by an external independent interview (Kiddie-SADS; Kaufman et al., 1996). The Kiddie-SADS interview will be conducted by a trained rater external to the project.
Change from baseline children´s psychiatric symptomatology at 48 months | baseline and 48 months
  Children´s psychiatric symptomatology will be assessed in all groups (intervention groups and control group) by an external independent interview (Kiddie-SADS; Kaufman et al., 1996). The Kiddie-SADS interview will be conducted by a trained rater external to the project.
Change from baseline children´s psychiatric symptomatology at 60 months | baseline and 60 months
  Children´s psychiatric symptomatology will be assessed in all groups (intervention groups and control group) by an external independent interview (Kiddie-SADS; Kaufman et al., 1996). The Kiddie-SADS interview will be conducted by a trained rater external to the project.

SECONDARY OUTCOMES:
Change from baseline children´s depressive symptomatology at 12 months | baseline and 12 months
  Children´s depressive symptomatology will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the "Children´s depression inventory" (Depressionsinventar für Kinder und Jugendliche (DIKJ); Stiensmeier-Pelster, Schürmann, & Duda, 2000).
  The German version of the "Children´s depression inventory" consists of 26 Items. Each item has 3 response options, which range from 0 = "symptom not present" to 2 = "symptom is very much present". The items are summed up to a total score (0-52), with higher values representing a higher number and more severe depressive symptoms.
Change from baseline children´s depressive symptomatology at 24 months | baseline and 24 months
  Children´s depressive symptomatology will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the "Children´s depression inventory" (Depressionsinventar für Kinder und Jugendliche (DIKJ); Stiensmeier-Pelster, Schürmann, & Duda, 2000).
  The German version of the "Children´s depression inventory" consists of 26 Items. Each item has 3 response options, which range from 0 = "symptom not present" to 2 = "symptom is very much present". The items are summed up to a total score (0-52), with higher values representing a higher number and more severe depressive symptoms.
Change from baseline children´s depressive symptomatology at 36 months | baseline and 36 months
  Children´s depressive symptomatology will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the "Children´s depression inventory" (Depressionsinventar für Kinder und Jugendliche (DIKJ); Stiensmeier-Pelster, Schürmann, & Duda, 2000).
  The German version of the "Children´s depression inventory" consists of 26 Items. Each item has 3 response options, which range from 0 = "symptom not present" to 2 = "symptom is very much present". The items are summed up to a total score (0-52), with higher values representing a higher number and more severe depressive symptoms.
Change from baseline children´s depressive symptomatology at 48 months | baseline and 48 months
  Children´s depressive symptomatology will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the "Children´s depression inventory" (Depressionsinventar für Kinder und Jugendliche (DIKJ); Stiensmeier-Pelster, Schürmann, & Duda, 2000).
  The German version of the "Children´s depression inventory" consists of 26 Items. Each item has 3 response options, which range from 0 = "symptom not present" to 2 = "symptom is very much present". The items are summed up to a total score (0-52), with higher values representing a higher number and more severe depressive symptoms.
Change from baseline children´s depressive symptomatology at 60 months | baseline and 60 months
  Children´s depressive symptomatology will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the "Children´s depression inventory" (Depressionsinventar für Kinder und Jugendliche (DIKJ); Stiensmeier-Pelster, Schürmann, & Duda, 2000).
  The German version of the "Children´s depression inventory" consists of 26 Items. Each item has 3 response options, which range from 0 = "symptom not present" to 2 = "symptom is very much present". The items are summed up to a total score (0-52), with higher values representing a higher number and more severe depressive symptoms.
Change from baseline children´s anxiety at 12 months | baseline and 12 months
  Children´s anxiety symptomatology will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the "Screen for child anxiety related emotional disorders" (Scared; Birmaher, Khetarpal, Cully, Brent, & McCanzie, 1995).
  The German version of the Scared consists of 41 items. Each item has 3 response options, which range from 0 = "not true or hardly ever true" to 2 = "true or often true". The subscales to be calculated are "panic/somatic" with a summed score ranging from 0 to 26, "generalized anxiety" with a summed score ranging from 0 to 18, "separation anxiety" with a summed score ranging from 0 to 16, "social phobia" with a summed score ranging from 0 to 14 and "school phobia" with a summed score ranging from 0 to 8. A total score can be obtained ranging from 0 to 82 by summing all scores. For all subscales and the total score higher values indicate a higher degree of anxiety.
Change from baseline children´s anxiety at 24 months | baseline and 24 months
  Children´s anxiety symptomatology will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the "Screen for child anxiety related emotional disorders" (Scared; Birmaher, Khetarpal, Cully, Brent, & McCanzie, 1995).
  The German version of the Scared consists of 41 items. Each item has 3 response options, which range from 0 = "not true or hardly ever true" to 2 = "true or often true". The subscales to be calculated are "panic/somatic" with a summed score ranging from 0 to 26, "generalized anxiety" with a summed score ranging from 0 to 18, "separation anxiety" with a summed score ranging from 0 to 16, "social phobia" with a summed score ranging from 0 to 14 and "school phobia" with a summed score ranging from 0 to 8. A total score can be obtained ranging from 0 to 82 by summing all scores. For all subscales and the total score higher values indicate a higher degree of anxiety.
Change from baseline children´s anxiety at 36 months | baseline and 36 months
  Children´s anxiety symptomatology will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the "Screen for child anxiety related emotional disorders" (Scared; Birmaher, Khetarpal, Cully, Brent, & McCanzie, 1995).
  The German version of the Scared consists of 41 items. Each item has 3 response options, which range from 0 = "not true or hardly ever true" to 2 = "true or often true". The subscales to be calculated are "panic/somatic" with a summed score ranging from 0 to 26, "generalized anxiety" with a summed score ranging from 0 to 18, "separation anxiety" with a summed score ranging from 0 to 16, "social phobia" with a summed score ranging from 0 to 14 and "school phobia" with a summed score ranging from 0 to 8. A total score can be obtained ranging from 0 to 82 by summing all scores. For all subscales and the total score higher values indicate a higher degree of anxiety.
Change from baseline children´s anxiety at 48 months | baseline and 48 months
  Children´s anxiety symptomatology will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the "Screen for child anxiety related emotional disorders" (Scared; Birmaher, Khetarpal, Cully, Brent, & McCanzie, 1995).
  The German version of the Scared consists of 41 items. Each item has 3 response options, which range from 0 = "not true or hardly ever true" to 2 = "true or often true". The subscales to be calculated are "panic/somatic" with a summed score ranging from 0 to 26, "generalized anxiety" with a summed score ranging from 0 to 18, "separation anxiety" with a summed score ranging from 0 to 16, "social phobia" with a summed score ranging from 0 to 14 and "school phobia" with a summed score ranging from 0 to 8. A total score can be obtained ranging from 0 to 82 by summing all scores. For all subscales and the total score higher values indicate a higher degree of anxiety.
Change from baseline children´s anxiety at 60 months | baseline and 60 months
  Children´s anxiety symptomatology will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the "Screen for child anxiety related emotional disorders" (Scared; Birmaher, Khetarpal, Cully, Brent, & McCanzie, 1995).
  The German version of the Scared consists of 41 items. Each item has 3 response options, which range from 0 = "not true or hardly ever true" to 2 = "true or often true". The subscales to be calculated are "panic/somatic" with a summed score ranging from 0 to 26, "generalized anxiety" with a summed score ranging from 0 to 18, "separation anxiety" with a summed score ranging from 0 to 16, "social phobia" with a summed score ranging from 0 to 14 and "school phobia" with a summed score ranging from 0 to 8. A total score can be obtained ranging from 0 to 82 by summing all scores. For all subscales and the total score higher values indicate a higher degree of anxiety.
Change from baseline parent reported children´s psychiatric symptoms at 12 months | baseline and 12 months
  Children´s psychiatric disorders will be assessed by parents´ rating of the German version of the "Child behavior checklist" (CBCL; Achenbach, 1991).
  The German version of the CBCL consists of 118 items. Each item has 3 response options, which range from 0 = "not true or seldom true" to 2 = "true or often true". The 8 syndrome scales to be calculated by summing are "social withdrawal" with scores ranging from 0 - 18, "physical discomfort" with scores ranging from 0 - 18, "anxiety/depression" with scores ranging from 0 - 28, "social difficulties" with scores ranging from 0 - 16, "schizoid/compulsive" scores ranging from 0 - 14, "attention deficits" with scores ranging from 0 - 22, "dissocial behavior" with scores ranging from 0 - 26, "aggressive behavior" with scores ranging from 0 - 40 and "other difficulties" with scores ranging from 0 - 66. A total score can be calculated by summing with scores ranging from 0 - 236. For all scales higher values indicate a higher problem level.
Change from baseline parent reported children´s psychiatric symptoms at 24 months | baseline and 24 months
  Children´s psychiatric disorders will be assessed by parents´ rating of the German version of the "Child behavior checklist" (CBCL; Achenbach, 1991).
  The German version of the CBCL consists of 118 items. Each item has 3 response options, which range from 0 = "not true or seldom true" to 2 = "true or often true". The 8 syndrome scales to be calculated by summing are "social withdrawal" with scores ranging from 0 - 18, "physical discomfort" with scores ranging from 0 - 18, "anxiety/depression" with scores ranging from 0 - 28, "social difficulties" with scores ranging from 0 - 16, "schizoid/compulsive" scores ranging from 0 - 14, "attention deficits" with scores ranging from 0 - 22, "dissocial behavior" with scores ranging from 0 - 26, "aggressive behavior" with scores ranging from 0 - 40 and "other difficulties" with scores ranging from 0 - 66. A total score can be calculated by summing with scores ranging from 0 - 236. For all scales higher values indicate a higher problem level.
Change from baseline parent reported children´s psychiatric symptoms at 36 months | baseline and 36 months
  Children´s psychiatric disorders will be assessed by parents´ rating of the German version of the "Child behavior checklist" (CBCL; Achenbach, 1991).
  The German version of the CBCL consists of 118 items. Each item has 3 response options, which range from 0 = "not true or seldom true" to 2 = "true or often true". The 8 syndrome scales to be calculated by summing are "social withdrawal" with scores ranging from 0 - 18, "physical discomfort" with scores ranging from 0 - 18, "anxiety/depression" with scores ranging from 0 - 28, "social difficulties" with scores ranging from 0 - 16, "schizoid/compulsive" scores ranging from 0 - 14, "attention deficits" with scores ranging from 0 - 22, "dissocial behavior" with scores ranging from 0 - 26, "aggressive behavior" with scores ranging from 0 - 40 and "other difficulties" with scores ranging from 0 - 66. A total score can be calculated by summing with scores ranging from 0 - 236. For all scales higher values indicate a higher problem level.
Change from baseline parent reported children´s psychiatric symptoms at 48 months | baseline and 48 months
  Children´s psychiatric disorders will be assessed by parents´ rating of the German version of the "Child behavior checklist" (CBCL; Achenbach, 1991).
  The German version of the CBCL consists of 118 items. Each item has 3 response options, which range from 0 = "not true or seldom true" to 2 = "true or often true". The 8 syndrome scales to be calculated by summing are "social withdrawal" with scores ranging from 0 - 18, "physical discomfort" with scores ranging from 0 - 18, "anxiety/depression" with scores ranging from 0 - 28, "social difficulties" with scores ranging from 0 - 16, "schizoid/compulsive" scores ranging from 0 - 14, "attention deficits" with scores ranging from 0 - 22, "dissocial behavior" with scores ranging from 0 - 26, "aggressive behavior" with scores ranging from 0 - 40 and "other difficulties" with scores ranging from 0 - 66. A total score can be calculated by summing with scores ranging from 0 - 236. For all scales higher values indicate a higher problem level.
Change from baseline parent reported children´s psychiatric symptoms at 60 months | baseline and 60 months
  Children´s psychiatric disorders will be assessed by parents´ rating of the German version of the "Child behavior checklist" (CBCL; Achenbach, 1991).
  The German version of the CBCL consists of 118 items. Each item has 3 response options, which range from 0 = "not true or seldom true" to 2 = "true or often true". The 8 syndrome scales to be calculated by summing are "social withdrawal" with scores ranging from 0 - 18, "physical discomfort" with scores ranging from 0 - 18, "anxiety/depression" with scores ranging from 0 - 28, "social difficulties" with scores ranging from 0 - 16, "schizoid/compulsive" scores ranging from 0 - 14, "attention deficits" with scores ranging from 0 - 22, "dissocial behavior" with scores ranging from 0 - 26, "aggressive behavior" with scores ranging from 0 - 40 and "other difficulties" with scores ranging from 0 - 66. A total score can be calculated by summing with scores ranging from 0 - 236. For all scales higher values indicate a higher problem level.
Change from baseline children´s self reported psychiatric symptoms at 12 months | baseline and 12 months
  Children´s psychiatric disorders will further be assessed by children´s rating of the German version of the "Youth self report" (YSR; Achenbach, 1991).
  The German version of the YSR consists of 119 items. Each item has 3 response options, which range from 0 = "not true or seldom true" to 2 = "true or often true". The 8 syndrome scales to be calculated by summing are "social withdrawal" with scores ranging from 0 - 14, "physical discomfort" with scores ranging from 0 - 18, "anxiety/depression" with scores ranging from 0 - 32, "social difficulties" with scores ranging from 0 - 16, "schizoid/compulsive" scores ranging from 0 - 14, "attention deficits" with scores ranging from 0 - 18, "dissocial behavior" with scores ranging from 0 - 22, "aggressive behavior" with scores ranging from 0 - 38 and "other difficulties" with scores ranging from 0 - 40. A total score can be calculated by summing with scores ranging from 0 - 238. For all scales higher values indicate a higher problem level.
Change from baseline children´s self reported psychiatric symptoms at 24 months | baseline and 24 months
  Children´s psychiatric disorders will further be assessed by children´s rating of the German version of the "Youth self report" (YSR; Achenbach, 1991).
  The German version of the YSR consists of 119 items. Each item has 3 response options, which range from 0 = "not true or seldom true" to 2 = "true or often true". The 8 syndrome scales to be calculated by summing are "social withdrawal" with scores ranging from 0 - 14, "physical discomfort" with scores ranging from 0 - 18, "anxiety/depression" with scores ranging from 0 - 32, "social difficulties" with scores ranging from 0 - 16, "schizoid/compulsive" scores ranging from 0 - 14, "attention deficits" with scores ranging from 0 - 18, "dissocial behavior" with scores ranging from 0 - 22, "aggressive behavior" with scores ranging from 0 - 38 and "other difficulties" with scores ranging from 0 - 40. A total score can be calculated by summing with scores ranging from 0 - 238. For all scales higher values indicate a higher problem level.
Change from baseline children´s self reported psychiatric symptoms at 36 months | baseline and 36 months
  Children´s psychiatric disorders will further be assessed by children´s rating of the German version of the "Youth self report" (YSR; Achenbach, 1991).
  The German version of the YSR consists of 119 items. Each item has 3 response options, which range from 0 = "not true or seldom true" to 2 = "true or often true". The 8 syndrome scales to be calculated by summing are "social withdrawal" with scores ranging from 0 - 14, "physical discomfort" with scores ranging from 0 - 18, "anxiety/depression" with scores ranging from 0 - 32, "social difficulties" with scores ranging from 0 - 16, "schizoid/compulsive" scores ranging from 0 - 14, "attention deficits" with scores ranging from 0 - 18, "dissocial behavior" with scores ranging from 0 - 22, "aggressive behavior" with scores ranging from 0 - 38 and "other difficulties" with scores ranging from 0 - 40. A total score can be calculated by summing with scores ranging from 0 - 238. For all scales higher values indicate a higher problem level.
Change from baseline children´s self reported psychiatric symptoms at 48 months | baseline and 48 months
  Children´s psychiatric disorders will further be assessed by children´s rating of the German version of the "Youth self report" (YSR; Achenbach, 1991).
  The German version of the YSR consists of 119 items. Each item has 3 response options, which range from 0 = "not true or seldom true" to 2 = "true or often true". The 8 syndrome scales to be calculated by summing are "social withdrawal" with scores ranging from 0 - 14, "physical discomfort" with scores ranging from 0 - 18, "anxiety/depression" with scores ranging from 0 - 32, "social difficulties" with scores ranging from 0 - 16, "schizoid/compulsive" scores ranging from 0 - 14, "attention deficits" with scores ranging from 0 - 18, "dissocial behavior" with scores ranging from 0 - 22, "aggressive behavior" with scores ranging from 0 - 38 and "other difficulties" with scores ranging from 0 - 40. A total score can be calculated by summing with scores ranging from 0 - 238. For all scales higher values indicate a higher problem level.
Change from baseline children´s self reported psychiatric symptoms at 60 months | baseline and 60 months
  Children´s psychiatric disorders will further be assessed by children´s rating of the German version of the "Youth self report" (YSR; Achenbach, 1991).
  The German version of the YSR consists of 119 items. Each item has 3 response options, which range from 0 = "not true or seldom true" to 2 = "true or often true". The 8 syndrome scales to be calculated by summing are "social withdrawal" with scores ranging from 0 - 14, "physical discomfort" with scores ranging from 0 - 18, "anxiety/depression" with scores ranging from 0 - 32, "social difficulties" with scores ranging from 0 - 16, "schizoid/compulsive" scores ranging from 0 - 14, "attention deficits" with scores ranging from 0 - 18, "dissocial behavior" with scores ranging from 0 - 22, "aggressive behavior" with scores ranging from 0 - 38 and "other difficulties" with scores ranging from 0 - 40. A total score can be calculated by summing with scores ranging from 0 - 238. For all scales higher values indicate a higher problem level.
Change from baseline children´s structural functioning at 12 months | baseline and 12 months
  Children´s structural functioning will be assessed by self-report (children and adolescents aged 10 years and older) using the German structure questionnaire for the "Operationalized psychodynamic diagnostic for children and adolescents" (OPD-KJ2-SF, Goth & Schmeck, 2016).
  The OPD-KJ2-SF consists of 81 items. Each item has 5 response options, which range from 0 = "no" to 4 = "yes". The 4 higher order scales to be calculated by summing are "self regulation" with scores ranging from 0 - 64, "identity" with scores ranging from 0 - 96, "interpersonality" with scores ranging from 0 - 100 and "attachment" with scores ranging from 0 - 64. A total score can be calculated ba summing with scores ranging from 0 - 342. For all scales higher values indicate a higher structural impairment.
Change from baseline children´s structural functioning at 24 months | baseline and 24 months
  Children´s structural functioning will be assessed by self-report (children and adolescents aged 10 years and older) using the German structure questionnaire for the "Operationalized psychodynamic diagnostic for children and adolescents" (OPD-KJ2-SF, Goth & Schmeck, 2017).
  The OPD-KJ2-SF consists of 81 items. Each item has 5 response options, which range from 0 = "no" to 4 = "yes". The 4 higher order scales to be calculated by summing are "self regulation" with scores ranging from 0 - 64, "identity" with scores ranging from 0 - 96, "interpersonality" with scores ranging from 0 - 100 and "attachment" with scores ranging from 0 - 64. A total score can be calculated ba summing with scores ranging from 0 - 342. For all scales higher values indicate a higher structural impairment.
Change from baseline children´s structural functioning at 36 months | baseline and 36 months
  Children´s structural functioning will be assessed by self-report (children and adolescents aged 10 years and older) using the German structure questionnaire for the "Operationalized psychodynamic diagnostic for children and adolescents" (OPD-KJ2-SF, Goth & Schmeck, 2017).
  The OPD-KJ2-SF consists of 81 items. Each item has 5 response options, which range from 0 = "no" to 4 = "yes". The 4 higher order scales to be calculated by summing are "self regulation" with scores ranging from 0 - 64, "identity" with scores ranging from 0 - 96, "interpersonality" with scores ranging from 0 - 100 and "attachment" with scores ranging from 0 - 64. A total score can be calculated ba summing with scores ranging from 0 - 342. For all scales higher values indicate a higher structural impairment.
Change from baseline children´s structural functioning at 48 months | baseline and 48 months
  Children´s structural functioning will be assessed by self-report (children and adolescents aged 10 years and older) using the German structure questionnaire for the "Operationalized psychodynamic diagnostic for children and adolescents" (OPD-KJ2-SF, Goth & Schmeck, 2017).
  The OPD-KJ2-SF consists of 81 items. Each item has 5 response options, which range from 0 = "no" to 4 = "yes". The 4 higher order scales to be calculated by summing are "self regulation" with scores ranging from 0 - 64, "identity" with scores ranging from 0 - 96, "interpersonality" with scores ranging from 0 - 100 and "attachment" with scores ranging from 0 - 64. A total score can be calculated ba summing with scores ranging from 0 - 342. For all scales higher values indicate a higher structural impairment.
Change from baseline children´s structural functioning at 60 months | baseline and 60 months
  Children´s structural functioning will be assessed by self-report (children and adolescents aged 10 years and older) using the German structure questionnaire for the "Operationalized psychodynamic diagnostic for children and adolescents" (OPD-KJ2-SF, Goth & Schmeck, 2017).
  The OPD-KJ2-SF consists of 81 items. Each item has 5 response options, which range from 0 = "no" to 4 = "yes". The 4 higher order scales to be calculated by summing are "self regulation" with scores ranging from 0 - 64, "identity" with scores ranging from 0 - 96, "interpersonality" with scores ranging from 0 - 100 and "attachment" with scores ranging from 0 - 64. A total score can be calculated ba summing with scores ranging from 0 - 342. For all scales higher values indicate a higher structural impairment.
Change from baseline children´s health related quality of life at 12 months | baseline and 12 months
  Children´s health related quality of life will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the Kidscreen-27 (Ravens-Sieberer & the European KIDSCREEN group, 2006).
  The Kidscreen-27 consists of 27 items. Each item is scored on a 5-point Likert scale ranging from 1 = "not at all true/never" to 5 = "extremely/always". The items are summed up for the 5 specific subscales "physical well-being" with scores ranging from 1 - 20, "psychological well-being" with scores ranging from 1 - 35, "autonomy and parent relation" with scores ranging from 1 - 35, "Social support and peers" with scores ranging from 1 - 40 and "school environment" with scores ranging from 1 - 20. High values represent a high quality of life.
Change from baseline children´s health related quality of life at 24 months | baseline and 24 months
  Children´s health related quality of life will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the Kidscreen-27 (Ravens-Sieberer & the European KIDSCREEN group, 2006).
  The Kidscreen-27 consists of 27 items. Each item is scored on a 5-point Likert scale ranging from 1 = "not at all true/never" to 5 = "extremely/always". The items are summed up for the 5 specific subscales "physical well-being" with scores ranging from 1 - 20, "psychological well-being" with scores ranging from 1 - 35, "autonomy and parent relation" with scores ranging from 1 - 35, "Social support and peers" with scores ranging from 1 - 40 and "school environment" with scores ranging from 1 - 20. High values represent a high quality of life.
Change from baseline children´s health related quality of life at 36 months | baseline and 36 months
  Children´s health related quality of life will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the Kidscreen-27 (Ravens-Sieberer & the European KIDSCREEN group, 2006).
  The Kidscreen-27 consists of 27 items. Each item is scored on a 5-point Likert scale ranging from 1 = "not at all true/never" to 5 = "extremely/always". The items are summed up for the 5 specific subscales "physical well-being" with scores ranging from 1 - 20, "psychological well-being" with scores ranging from 1 - 35, "autonomy and parent relation" with scores ranging from 1 - 35, "Social support and peers" with scores ranging from 1 - 40 and "school environment" with scores ranging from 1 - 20. High values represent a high quality of life.
Change from baseline children´s health related quality of life at 48 months | baseline and 48 months
  Children´s health related quality of life will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the Kidscreen-27 (Ravens-Sieberer & the European KIDSCREEN group, 2006).
  The Kidscreen-27 consists of 27 items. Each item is scored on a 5-point Likert scale ranging from 1 = "not at all true/never" to 5 = "extremely/always". The items are summed up for the 5 specific subscales "physical well-being" with scores ranging from 1 - 20, "psychological well-being" with scores ranging from 1 - 35, "autonomy and parent relation" with scores ranging from 1 - 35, "Social support and peers" with scores ranging from 1 - 40 and "school environment" with scores ranging from 1 - 20. High values represent a high quality of life.
Change from baseline children´s health related quality of life at 60 months | baseline and 60 months
  Children´s health related quality of life will be assessed by children´s (aged 10 years and older) and parents´ rating of the German version of the Kidscreen-27 (Ravens-Sieberer & the European KIDSCREEN group, 2006).
  The Kidscreen-27 consists of 27 items. Each item is scored on a 5-point Likert scale ranging from 1 = "not at all true/never" to 5 = "extremely/always". The items are summed up for the 5 specific subscales "physical well-being" with scores ranging from 1 - 20, "psychological well-being" with scores ranging from 1 - 35, "autonomy and parent relation" with scores ranging from 1 - 35, "Social support and peers" with scores ranging from 1 - 40 and "school environment" with scores ranging from 1 - 20. High values represent a high quality of life.
Change from baseline children´s global impairment at 12 months | baseline and 12 months
  Children´s global impairment will be assessed by a trained rater external to the project using the german "Skala zur Gesamtbeurteilung von Kindern und Jugendlichen" (SGKJ; Steinhausen, 1985).
  The SGKJ is a 10 point scale which describes a hypothetic continuum from 10 = mental health ("Outstanding functioning in all areas - e.g. at home, in school, with peers") to 1 = mental disorder ("Needs steady supervision because of severe aggressive or self-destructive behavior, impaired reality testing, communication, cognition, affect or hygiene").
Change from baseline children´s global impairment at 24 months | baseline and 24 months
  Children´s global impairment will be assessed by a trained rater external to the project using the german "Skala zur Gesamtbeurteilung von Kindern und Jugendlichen" (SGKJ; Steinhausen, 1985).
  The SGKJ is a 10 point scale which describes a hypothetic continuum from 10 = mental health ("Outstanding functioning in all areas - e.g. at home, in school, with peers") to 1 = mental disorder ("Needs steady supervision because of severe aggressive or self-destructive behavior, impaired reality testing, communication, cognition, affect or hygiene").
Change from baseline children´s global impairment at 36 months | baseline and 36 months
  Children´s global impairment will be assessed by a trained rater external to the project using the german "Skala zur Gesamtbeurteilung von Kindern und Jugendlichen" (SGKJ; Steinhausen, 1985).
  The SGKJ is a 10 point scale which describes a hypothetic continuum from 10 = mental health ("Outstanding functioning in all areas - e.g. at home, in school, with peers") to 1 = mental disorder ("Needs steady supervision because of severe aggressive or self-destructive behavior, impaired reality testing, communication, cognition, affect or hygiene").
Change from baseline children´s global impairment at 48 months | baseline and 48 months
  Children´s global impairment will be assessed by a trained rater external to the project using the german "Skala zur Gesamtbeurteilung von Kindern und Jugendlichen" (SGKJ; Steinhausen, 1985).
  The SGKJ is a 10 point scale which describes a hypothetic continuum from 10 = mental health ("Outstanding functioning in all areas - e.g. at home, in school, with peers") to 1 = mental disorder ("Needs steady supervision because of severe aggressive or self-destructive behavior, impaired reality testing, communication, cognition, affect or hygiene").
Change from baseline children´s global impairment at 60 months | baseline and 60 months
  Children´s global impairment will be assessed by a trained rater external to the project using the german "Skala zur Gesamtbeurteilung von Kindern und Jugendlichen" (SGKJ; Steinhausen, 1985).
  The SGKJ is a 10 point scale which describes a hypothetic continuum from 10 = mental health ("Outstanding functioning in all areas - e.g. at home, in school, with peers") to 1 = mental disorder ("Needs steady supervision because of severe aggressive or self-destructive behavior, impaired reality testing, communication, cognition, affect or hygiene").
Change from baseline relational functioning at 12 months | baseline and 12 months
  Families´ relational functioning will be rated by a trained rater external to the project using the german version of the "Global assessment of relational functioning scale" (GARF; Saß, Wittchen, & Zaudig, 1996).
  The GARF is a 100 point continuous scale with anchor items for every 20 points. It assesses the family functioning from 1 -20 = "the system of relationships within the family is extremely disturbed, continuity of contact and attachment can not be kept up any longer" to 80 - 100 = "the system of relationships in the family ist high functioning".
Change from baseline relational functioning at 24 months | baseline and 24 months
  Families´ relational functioning will be rated by a trained rater external to the project using the german version of the "Global assessment of relational functioning scale" (GARF; Saß, Wittchen, & Zaudig, 1996).
  The GARF is a 100 point continuous scale with anchor items for every 20 points. It assesses the family functioning from 1 -20 = "the system of relationships within the family is extremely disturbed, continuity of contact and attachment can not be kept up any longer" to 80 - 100 = "the system of relationships in the family ist high functioning".
Change from baseline relational functioning at 36 months | baseline and 36 months
  Families´ relational functioning will be rated by a trained rater external to the project using the german version of the "Global assessment of relational functioning scale" (GARF; Saß, Wittchen, & Zaudig, 1996).
  The GARF is a 100 point continuous scale with anchor items for every 20 points. It assesses the family functioning from 1 -20 = "the system of relationships within the family is extremely disturbed, continuity of contact and attachment can not be kept up any longer" to 80 - 100 = "the system of relationships in the family ist high functioning".
Change from baseline relational functioning at 48 months | baseline and 48 months
  Families´ relational functioning will be rated by a trained rater external to the project using the german version of the "Global assessment of relational functioning scale" (GARF; Saß, Wittchen, & Zaudig, 1996).
  The GARF is a 100 point continuous scale with anchor items for every 20 points. It assesses the family functioning from 1 -20 = "the system of relationships within the family is extremely disturbed, continuity of contact and attachment can not be kept up any longer" to 80 - 100 = "the system of relationships in the family ist high functioning".
Change from baseline relational functioning at 60 months | baseline and 60 months
  Families´ relational functioning will be rated by a trained rater external to the project using the german version of the "Global assessment of relational functioning scale" (GARF; Saß, Wittchen, & Zaudig, 1996).
  The GARF is a 100 point continuous scale with anchor items for every 20 points. It assesses the family functioning from 1 -20 = "the system of relationships within the family is extremely disturbed, continuity of contact and attachment can not be kept up any longer" to 80 - 100 = "the system of relationships in the family ist high functioning".
Change from baseline children´s global functioning at 12 months | baseline and 12 months
  Children´s global functioning will be rated by a trained rater external to the project using the german version of the "Global assessment functioning scale" (GAF; American Psychiatric Association, 2000).
  The GAF is a 100 point continuous scale with anchor items for every 10 points. Scores between 91 - 100 are given for "Outstanding performance in many activities and coping, no loss of control, being appreciated for many positive qualities, no symptoms". Scores between 1 - 10 are given for "permanent danger of hurting self or others or persistent inability to maintain minimal personal hygiene or serious suicidal attempt with clear expectation of death".
Change from baseline children´s global functioning at 24 months | baseline and 24 months
  Children´s global functioning will be rated by a trained rater external to the project using the german version of the "Global assessment functioning scale" (GAF; American Psychiatric Association, 2000).
  The GAF is a 100 point continuous scale with anchor items for every 10 points. Scores between 91 - 100 are given for "Outstanding performance in many activities and coping, no loss of control, being appreciated for many positive qualities, no symptoms". Scores between 1 - 10 are given for "permanent danger of hurting self or others or persistent inability to maintain minimal personal hygiene or serious suicidal attempt with clear expectation of death".
Change from baseline children´s global functioning at 36 months | baseline and 36 months
  Children´s global functioning will be rated by a trained rater external to the project using the german version of the "Global assessment functioning scale" (GAF; American Psychiatric Association, 2000).
  The GAF is a 100 point continuous scale with anchor items for every 10 points. Scores between 91 - 100 are given for "Outstanding performance in many activities and coping, no loss of control, being appreciated for many positive qualities, no symptoms". Scores between 1 - 10 are given for "permanent danger of hurting self or others or persistent inability to maintain minimal personal hygiene or serious suicidal attempt with clear expectation of death".
Change from baseline children´s global functioning at 48 months | baseline and 48 months
  Children´s global functioning will be rated by a trained rater external to the project using the german version of the "Global assessment functioning scale" (GAF; American Psychiatric Association, 2000).
  The GAF is a 100 point continuous scale with anchor items for every 10 points. Scores between 91 - 100 are given for "Outstanding performance in many activities and coping, no loss of control, being appreciated for many positive qualities, no symptoms". Scores between 1 - 10 are given for "permanent danger of hurting self or others or persistent inability to maintain minimal personal hygiene or serious suicidal attempt with clear expectation of death".
Change from baseline children´s global functioning at 60 months | baseline and 60 months
  Children´s global functioning will be rated by a trained rater external to the project using the german version of the "Global assessment functioning scale" (GAF; American Psychiatric Association, 2000).
  The GAF is a 100 point continuous scale with anchor items for every 10 points. Scores between 91 - 100 are given for "Outstanding performance in many activities and coping, no loss of control, being appreciated for many positive qualities, no symptoms". Scores between 1 - 10 are given for "permanent danger of hurting self or others or persistent inability to maintain minimal personal hygiene or serious suicidal attempt with clear expectation of death".
Change from baseline health economic data at 12 months | baseline and 12 months
  Health economics will be assessed by a trained rater external to the project using the german version of the "Children and adolescent mental health services receipt inventory" (CAMHSRI-DE; Kilian et al., 2009).
  The CAMHSRI-DE assesses demand (number and duration) of inpatient and outpatient medical services as well as use of medication and demand of special educational establishment or offers in school in the past 12 months.
Change from baseline health economic data at 24 months | baseline and 24 months
  Health economics will be assessed by a trained rater external to the project using the german version of the "Children and adolescent mental health services receipt inventory" (CAMHSRI-DE; Kilian et al., 2009).
  The CAMHSRI-DE assesses demand (number and duration) of inpatient and outpatient medical services as well as use of medication and demand of special educational establishment or offers in school in the past 12 months.
Change from baseline health economic data at 36 months | baseline and 36 months
  Health economics will be assessed by a trained rater external to the project using the german version of the "Children and adolescent mental health services receipt inventory" (CAMHSRI-DE; Kilian et al., 2009).
  The CAMHSRI-DE assesses demand (number and duration) of inpatient and outpatient medical services as well as use of medication and demand of special educational establishment or offers in school in the past 12 months.
Change from baseline health economic data at 48 months | baseline and 48 months
  Health economics will be assessed by a trained rater external to the project using the german version of the "Children and adolescent mental health services receipt inventory" (CAMHSRI-DE; Kilian et al., 2009).
  The CAMHSRI-DE assesses demand (number and duration) of inpatient and outpatient medical services as well as use of medication and demand of special educational establishment or offers in school in the past 12 months.
Change from baseline health economic data at 60 months | baseline and 60 months
  Health economics will be assessed by a trained rater external to the project using the german version of the "Children and adolescent mental health services receipt inventory" (CAMHSRI-DE; Kilian et al., 2009).
  The CAMHSRI-DE assesses demand (number and duration) of inpatient and outpatient medical services as well as use of medication and demand of special educational establishment or offers in school in the past 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Silke Wiegand-Grefe, Prof. Dr., Principal Investigator — UKE Universitätsklinikum Hamburg-Eppendorf